CLINICAL TRIAL: NCT06181916
Title: Quantitative and Qualitative Research for "A Video-Based Mobile Health Program to Support People Living With HIV Across the HIV Care Continuum"
Brief Title: Quantitative and Qualitative Research for "mHealth Program to Support People Living With HIV Across the HIV Care Continuum"
Acronym: VSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sentient Research (Industry)
Collaborators: AIDS Healthcare Foundation (Other); Los Angeles LGBT Center (Other); University of Mississippi Medical Center (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9043
Record Dates: First submitted 2023-12-02; First posted 2023-12-26 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
Keywords: HIV; mHealth; viral load; HIV disparities; HIV care continuum
MeSH Terms: conditions — HIV Infections | interventions — Adenosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amp mHealth App (Experimental): Amp, video-based, virtual support system on an mHealth platform with resources and tools to help YBMSM living with HIV become and stay virally suppressed.
  Interventions: Behavioral: Amp
- Standard of Care (No Intervention): Standard of care (SOS) linkage to care services typically provided by linkage specialists, health navigators, or case workers.

INTERVENTIONS:
Behavioral: Amp — Amp is a virtual support system mHealth app that provides information and social support to help young Black men who have sex with men (YBMSM) living with HIV achieve better HIV care continuum outcomes and overall well-being.
  Arms: Amp mHealth App

SUMMARY:
The goal of this randomized control trial (RCT) is to assess the effectiveness of Amp, a mobile health (mHealth) app designed to improve outcomes along the HIV care continuum for young Black men who have sex with men (YBMSM) living with HIV. HIV care continuum (linkage to care, retention, viral suppression), quality of life and self efficacy outcomes will be compared after a 4-month period between the intervention group (use Amp and standard of care) and the control group (standard of care only).

DETAILED DESCRIPTION:
A maximum of 400 YBMSM participants will be recruited into a randomized control trial from multiple sites across the US to assess the effectiveness of Amp, an mHealth app designed to improve outcomes along the HIV care continuum for YBMSM living with HIV. HIV care continuum (linkage to care, retention, viral suppression), quality of life and self efficacy outcomes will be compared after a 4-month period between the intervention group (use Amp and standard of care) and the control group (standard of care only).

ELIGIBILITY:
Inclusion Criteria:

* MSM AND;
* Black or African-American AND;
* 18-29 years old AND;
* Diagnosed with HIV during the study period (From April 1, 2024-August 31 2024) OR;
* Diagnosed with HIV in the year prior to the study period (April 1, 2023-March 31, 2024) OR;
* HIV positive but not linked into care OR;
* Fallen out of care (no HIV care visits within last 6 months) OR;
* Currently in care but NOT virally suppressed (viral load ≥200 copies/mL)
* AND, Online access through a mobile device AND;
* Ability to read and write English.

Exclusion Criteria:

* Currently participating in another HIV care continuum or mobile health intervention
* Plan to leave the study site within the study period
* Cognitively impaired at recruitment or baseline testing
* Has a self-reported health issue that prohibits them from participating

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 4 months
  HIV viral load is less than 200 copies per microliter based on labs in patient EMR data. Viral suppression (viral load is less than 200 copies per microliter) is the better outcome.
HIV Stigma | 4 months
  Composite agreement score on 13 HIV related stigma statements as measured by items derived from the Berger HIV Stigma Scale. Agreement from 1 (Strongly Disagree) to 5 (Strongly Agree). Lower scores indicate lower stigma (better outcome). Range of composite scores will be from 13 to 65.

SECONDARY OUTCOMES:
HIV and Anti-retroviral knowledge | 4 months
  Composite agreement score on 7 knowledge statements around Anti-retroviral, viral suppression, and U=U. Agreement from 1 (Strongly Disagree) to 5 (Strongly Agree). Higher scores indicate greater knowledge (better outcome). Range of composite scores will be from 7 to 35.
Anti-retroviral medication adherence | 4 months
  Self-report measures of ART adherence based on type of prescription (injectable or pill), length of time taking medication, and time since last does in moths and/or days.
Adherence barriers | 4 months
  Reasons checked for not taking ART medication from a list of 13 reasons and an "other" write in. More reasons checked indicate more barriers. Little to no barriers is the better outcome. Composite score range for reasons is from 0 to 13. A lower score is the better outcome.
Self-Reported Medical Visits | 4 months
  Self-reported completed medical visits and appointments missed in the past 4 months. Response range is from "0" to "30 or more times". A lower selection is the better outcome.
HIV status disclosure | 4 months
  Self report measures of HIV status disclosure.
Social support | 4 months
  Composite agreement score on 7 statements for social support. Agreement from 1 (Strongly Disagree) to 5 (Strongly Agree). Higher scores indicate higher social support (better outcome). Range of composite scores will be from 7 to 35.
Depressive symptoms | 4 months
  Composite frequency score on 6 depression symptoms from the Brief Symptom Inventory 18 (BSI-18). From 1 (Not at all) to 4 (Nearly every day). Lower scores indicate lower frequency of symptoms (better outcome). Range of composite scores will be from 6 to 24.
Anxiety symptoms | 4 months
  Composite frequency score on 5 anxiety symptoms from the Brief Symptom Inventory 18 (BSI-18). From 1 (Not at all) to 4 (Nearly every day). Lower scores indicate lower frequency of symptoms (better outcome). Range of composite scores will be from 5 to 20.
Substance use | 4 months
  Composite score on self-report measures of substance use for 10 substances and an "other" write-in from 1 (Never) to 5 (Every day). Range of scores from 10 to 55. A lower score is the better outcome.
Time to Treatment Initiation | 4 months
  Time in days to treatment initiation from date of diagnosis or referral.
Linkage to HIV Care | 4 months
  Linkage to HIV care based on two completed medical visits from date of diagnosis or referral.
Medical Visits Record based on EMR | 4 months
  Completed medical visits and appointments missed in the past 4 months based on electronic medical record.
HIV Self-Management | 4 months
  Composite agreement score on 12 HIV self-management agreement statements. Agreement from 1 (Strongly Disagree) to 5 (Strongly Agree). Lower scores indicate lower self-management and higher scores indicate higher HIV self-management stigma (better outcome). Range of composite scores will be from 12 to 60.
Resilience | 4 months
  Composite agreement score on resilience agreement statements. Agreement from 1 (Strongly Disagree) to 5 (Strongly Agree). Lower scores indicate lower resilience and higher scores indicate higher resilience (better outcome). Range of composite score from 8 to 40.
Discussion of PrEP with Sex Partners | 4 months
  Frequency on a 5-point scale from "never" to "all of the time" on discussing PrEP with an HIV negative or unknown status partner in the last 4 months.
Discussion of U=U with Sex Partners | 4 months
  Frequency on a 5-point scale from "never" to "all of the time" on discussing U=U with an HIV negative or unknown status partner in the last 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Montoya, PhD, Principal Investigator — Sentient Research
Locations (1):
- Sentient Research, West Covina, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is currently undecided.